CLINICAL TRIAL: NCT05960994
Title: Evaluation of the Clinical Impact of Different Telemedicine Practices in Intensive Care Units: a Stepped-wedge Cluster Randomized Clinical Trial
Brief Title: Evaluation of the Clinical Impact of Different Telemedicine Practices in Intensive Care Units
Acronym: Telescope_2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 5535-23
Record Dates: First submitted 2023-06-30; First posted 2023-07-27 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-06

CONDITIONS: Telemedicine; Critical Care; Intensive Care Units
Keywords: Telemedicine; Critical care; Intensive care units

STUDY DESIGN:
Intervention Model Description: The TELESCOPE II study is an open-label, national, multicenter, stepped-wedge cluster randomized controlled trial. The randomization unit will be the ICU, since the intervention will be applied to the entire multiprofessional team. Therefore, 25 ICUs participating in the study will be allocated and randomized to one of the five sequences. In each sequence, the initial period will serve as the control period without any intervention. Subsequently, as the intervention is stepwise implemented, new control periods will be introduced based on the assigned sequence. Due to the multifaceted nature of the intervention, a delay in onset of effect is expected; thus, the study design contemplates a transition period, which will occur in all sequences, when the intervention will be occurring, but these data will not be used in the main analysis. All groups will receive all interventions, but at different times
Masking Description: For technical reasons, it is impossible to perform blinding for patients, health care staff, professionals involved in patient care, and data collectors in the ICUs participating in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sequence 1 (Experimental): Sequence 1 will consist of a 3-month control period, followed by a 3-month transition period, and finally, a 19-month intervention period. The total duration of sequence 1 will be 25 months.
  Interventions: Other: Intervention period
- Sequence 2 (Experimental): Sequence 2 will consist of a 7-month control period, followed by a 3-month transition period, and finally, a 15-month intervention period. The total duration of sequence 2 will be 25 months.
  Interventions: Other: Intervention period
- Sequence 3 (Experimental): Sequence 3 will consist of a 11-month control period, followed by a 3-month transition period, and finally, a 9-month intervention period. The total duration of sequence 3 will be 25 months.
  Interventions: Other: Intervention period
- Sequence 4 (Experimental): Sequence 4 will consist of a 15-month control period, followed by a 3-month transition period, and finally, a 7-month intervention period. The total duration of sequence 4 will be 25 months.
  Interventions: Other: Intervention period
- Sequence 5 (Experimental): Sequence 5 will consist of a 19-month control period, followed by a 3-month transition period, and finally, a 3-month intervention period. The total duration of sequence 5 will be 25 months.
  Interventions: Other: Intervention period

INTERVENTIONS:
Other: Intervention period — During the intervention period, three interventions will be implemented through telemedicine.
  1. A daily multidisciplinary round conducted by a physician specialized in intensive care medicine.
  2. A intervention package administered by a specialized multidisciplinary team, consisting of nursing, physiotherapy, and clinical pharmacy.
  3. A management intervention package will be implemented, with a specific focus on enhancing quality and safety.

SUMMARY:
The objective of this study is to assess whether an intervention package via telemedicine consisting of daily multidisciplinary rounds with a specialist in intensive care medicine, an intervention package provided by a specialized multiprofessional team (nursing, physical therapy and clinical pharmacy) and a management intervention package, focused on quality and safety, reduces the length of stay in ICU patients in Brazil. Our hypothesis is that the intervention package via telemedicine has the potential to decrease the length of stay in ICU patients in Brazil.

The study provides for the implementation of three interventions in association via telemedicine.

* Daily multidisciplinary rounds conducted by a physician specialized in intensive care medicine
* Intervention package by specialized multidisciplinary team (nursing, physiotherapy and clinical pharmacy).
* Management intervention package (quality and safety).

The main questions it aims to answer are:

* Length of stay in ICU, measured in days, considering the time interval between admission to the ICU and the moment of physical transfer of the patient to another hospital admission area or external transfer.
* ICU mortality.
* Mechanical ventilation free time at 28 days.
* Ventilator-associated events.
* Patient Mobilization Density.
* Standard resource use.
* Standardized mortality rate.

DETAILED DESCRIPTION:
BACKGROUND:

ICU beds represent a scarce and high cost resource. This scenario is aggravated by the scarcity and heterogeneous distribution of specialists in intensive care medicine in Brazil. Telemedicine is an innovative and promising technology, with the possibility of making the daily multidisciplinary round accessible with the presence of intensive care medicine specialists throughout the national territory. In a previous study (Telescope Trial I), it was demonstrated that daily multidisciplinary round conducted via telemedicine by a remotely located medical specialist is a safe and feasible practice. However, little is known about different modalities of telemedicine care in the ICU environment, more specifically, about the impact of interventions performed by a multidisciplinary team (non-medical) and management interventions (quality and safety).

SAMPLE SIZE CALCULATION:

A total sample size of 18,750 to 25,000 patients will be considered to detect a reduction in the length of stay in the ICU on a logarithmic scale of 0.1479 (equivalent to a 1.1-day reduction compared to the baseline), resulting from the intervention package with a significance level of 5% and a minimum power of 95%. This variation in total sample size is due to different estimates of patients per period in the 25 Brazilian ICUs in question. It is estimated that there will be a variation of 30 to 40 patients recruited per month per ICU.

PRIMARY OUTCOME:

Length of stay in the ICU, measured in days, considering the time interval between admission to the ICU and the moment of physical transfer of the patient to another hospital admission area or external transfer.

SECONDARY OUTCOMES:

* ICU mortality.
* Mechanical ventilation free time in 28 days.
* Ventilator-associated events.
* Patient Mobilization Density.
* Standard resource use.
* Standardized mortality rate.

EXPLORATORY OUTCOMES:

* In-hospital mortality.
* Adherence to elevated bedside.
* Adequate prevention of venous thromboembolism.
* Accidental extubation rate.
* Rate of patients with adequate glycemic control (defined as blood glucose <70mg/dl to >180mg/dl).
* Rate of patients - day receiving oral or enteral diet.
* Rate of patient-day under adequate sedation [defined by Richmond agitation and sedation scale (RASS) = -3 to +].
* Rate of patients on oxygen therapy in normoxia [defined as peripheral oxygen saturation (SpO2) ≤92% to ≥96%].
* Rate of ICU readmission within 48 hours.
* Rate of early reintubation (<48h after extubation).
* Rate of central venous catheter use.
* Rate of indwelling urinary catheter use.
* Central venous catheter use time.
* Time of indwelling urinary catheter use.

STATISTICAL ANALYSIS:

All analyses will be described in detail in a statistical analysis plan, which will be finalized and submitted for publication before the database is closed and analyses begin. The primary statistical analyses will be conducted according to the intention-to-treat principle. Since ICUs will be randomized (not patients) and outcomes will be measured at the patient level, all analyses will be adjusted for clustering of data.

The primary outcome, length of ICU stay, will be analyzed at the individual level using a generalized linear mixed model, including as fixed effect the group, and considering distributions that can fit an expected right skewness (such as truncated Poisson, Gamma or inverse Gaussian distribution, etc.), choosing the best fit according to model parameters. The goal of the mixed model is to be able to fit random vectors, taking into account the correlation of the observations of individuals in the same cluster. Thus, the model will have as random effect an intercept for each unit. To consider an eventual lack of balance, we will adjust the analysis model for the factors used in the stratification and for the outcome value at the unit level in the pre-randomization period (i.e., mean length of stay in the ICU of each unit), as suggested by the literature. Additionally, we will adjust for factors that have a correlation with length of stay, aiming to decrease variability between units, thus impacting intra cluster correlation and increasing the power of the study. The adjustment factors will be defined after the pre-randomization period data collection, and reported in a statistical analysis plan, published before closing the study database, as specified above. These factors are about severity (SAPS 3) and clinical or surgical profile. In the event of a significant amount of missing data on the primary endpoint, the analysis will be re-evaluated after using multiple imputation with chained equations, assuming that the data will be missing at random. Data collected during the transition period will not be analyzed for primary, secondary or exploratory endpoints.

Sensitivity analyses and subgroups for the primary outcome:

We will define, a priori, the following subgroups for analysis of the primary outcome:

A - ICU length of stay stratified by clinical vs elective surgical and emergency surgical patients.

B - Length of stay in ICU stratified by three groups (lower, middle and upper thirds) of severity determined by SAPS 3 score.

C - ICU length of stay stratified by mechanically ventilated patients on admission (invasive mechanical ventilation).

Similarly, in all other analyses, generalized linear mixed models will be used. Analyses of the pre-specified secondary outcomes and subgroup analyses will not be adjusted for multiple comparisons, thus should be interpreted as exploratory.

Due to the importance of the SAPS 3 severity score, we will evaluate the calibration of the model with data from the pre-randomization period. If necessary, we will recalibrate the model for the study population.

The significance level for all endpoints will be 0.05. All analyses will be performed with R software (version 4.2.0, the version will be updated at the time of the analysis).

REGULATORY STATUS:

The study will be conducted in accordance with the principles of the Declaration of Helsinki and in accordance with the Medical Research Involving Humans Act.

APPROVAL FROM ETHICS AND REGULATORY AUTHORITIES:

The study will be performed according to the national and international guidelines. The Institutional Review Board of the Hospital Israelita Albert Einstein has approved this study (CAAE: 69575123.0.1001.0071). The participating centers will not initiate the study until they have obtained approval from their respective local Institutional Review Boards. The need for informed consent is determined by the Institutional Review Board of each participating center.

ELIGIBILITY:
Inclusion Criteria for Intensive care units:

* Intensive care units from public or philanthropic hospitals.
* Intensive care units with physician and nurses available 24 hours a day and physiotherapist available at least ≥ 18 hours a day.

Exclusion Criteria for Intensive care units:

* Intensive care units with structured multidisciplinary round more than three times a week conducted by an intensive care physician (certified), documented in the medical record, with a fixed duration (>5 min / patient), using some supporting tool (checklist or standard form), goal oriented, based on established protocols, including all the patients admitted to the ICU.
* Intensive care units already doing audit and feedback with specific planning.
* Dedicated coronary care units/cardiac intensive care units or other specialized units (cardiac surgery, neurological, burned patients).
* Step-down units or semi-intensive cardiac care unit.
* Intensive care units without availability of substitute renal therapy.
* ICU coordinator specialist in intensive care medicine and management training (MBA in Health Management or equivalent).

Inclusion Criteria for patients:

* Adult patients (≥ 18 years old).

Exclusion Criteria for patients:

* Admission for other reasons than medical (e.g., judicial cause, legal reasons, safety reasons).
* Previously included in the TELESCOPE II trial (for the primary outcome analysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25000 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Unit Length of Stay | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Time until discharge from the intensive care unit

SECONDARY OUTCOMES:
Mortality in the Intensive Care Unit | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Any death during Intensive Care Unit stay
Ventilator-free days at day 28 | 28 Days
  Number od days if the patient was extubated before 28 days and remained alive at day 28. Ventilator-free days at 28 days was the day between extubation and day 28. If the patient dies or remains intubated within 28 days, the patient is awarded zero actual Ventilator-free days at 28 days. The outcome does not indicate if the patient was re-intubated or died within 28 days after being extubated.
Ventilator-associated events | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Following the Centers for Disease Control and Prevention (CDC) 2013
Patient Mobilization Density | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Density of mobilization activities performed.
Standard resource use | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Calculated based on length of stay in the intensive care unit and adjusted for severity of acute illness
Standard mortality rate | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Ratio of observed deaths to expected deaths

OTHER OUTCOMES:
In-hospital mortality | From date of randomization until the date of hospital discharge or death, whichever comes first, assessed up to 90 days
  Any death during hospital stay
Rate of Patients with Head of the Bed Elevated | 30-45 degrees in patients under mechanical ventilation
  From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
Standard hospital mortality rate | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Ratio of observed hospital deaths to expected hospital deaths
Rate of adequate prophylaxis for venous thromboembolism | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Adequate prophylaxis for venous thromboembolism
Rate of adequate glycemic control | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Adequate glycemic control
Patient-days receiving oral or enteral feeding | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Use of enteral or oral feeding
Patient-days under light sedation or alert and calm | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Defined as a Richmond Agitation-Sedation Scale (RASS) -3 to +1
Rate of patients under normoxia | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Defined as oxygen saturation (SpO2) between 92% and 96%
Intensive care unit readmission | From date of randomization until the date of hospital discharge or death, whichever comes first, assessed up to 90 days
  Readmission less than 48 hours after discharge
Incidence of early reintubation | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Less than 48 hours after extubation
Rate of central-line catheter use | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Use of central-line catheter use
Rate of vesical catheter use | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Use of vesical catheter
Duration of central line catheter use | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Duration in days of central line catheter use
Duration of vesical catheter use | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Duration in days of vesical catheter use
Rate of daily multidisciplinary rounds performed | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Daily multidisciplinary rounds performed
Rate of recommendations performed, accepted and not validated / daily multidisciplinary rounds. | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  recommendations performed during the daily multidisciplinary rounds accepted and not validated

CONTACTS AND LOCATIONS:
Overall Officials: Adriano J Pereira, MD, PhD., Study Director — Hospital Israelita Albert Einstein; Renato CF Chaves, MD, MBA., Principal Investigator — Hospital Israelita Albert Einstein

IPD SHARING:
Plan to Share IPD: Yes
Data sharing open to researchers not members of the study after two years of the publication of the main study.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After two years of the first publication
Access Criteria: Data will be accessed through an online repository protected with password and for secondary analyses according to pre-specified plans.